CLINICAL TRIAL: NCT04056741
Title: A Supraglottic Instillation Device for Administration of Surfactant in Neonates- A Pilot Study
Brief Title: Administration of Surfactant Through an Instillation Device Infasurf® (Calfactant) in Neonates- A Pilot Study
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: alteration of study required
Sponsor: ONY (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ProVia-01
Record Dates: First submitted 2019-08-06; First posted 2019-08-14 (Actual); Last update posted 2023-11-01 (Actual); Status verified 2023-10

CONDITIONS: RDS of Prematurity; Surfactant Protein B Deficiency; Chronic Lung Disease
Keywords: Neonatal RDS; RDS; Surfactant Deficiency
MeSH Terms: conditions — Respiratory Distress Syndrome In Premature Infants; Surfactant Metabolism Dysfunction, Pulmonary, 1

STUDY DESIGN:
Intervention Model Description: Pilot Study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Surfactant administered via supraglottic administration device (Experimental): Patients in this group will have Calfactant at 3ml/kg administered via the supraglottic administration device.
  Interventions: Combination Product: surfactant airway device

INTERVENTIONS:
Combination Product: surfactant airway device — Infants who meet eligibility criteria and have a signed consent form by their parent or guardian will be enrolled in the study. Once enrolled, the surfactant airway device placement and surfactant administration will occur as detailed in the protocol. The infant will be monitored. If the infant meets instillation failure criteria, the procedure will be repeated shortly after the initial procedure. A maximum of two (2) doses will be given during the initial procedure. If the infant meets re-dosing criteria, (s)he may receive up to two (2) additional doses through the surfactant airway device (initial procedure with 1-2 doses and up to two additional doses). If at any time the infant reaches treatment failure criteria, the infant would be intubated and receive a site-specific surfactant through an endotracheal tube. Study outcome data will be followed until discharge from the NICU.

SUMMARY:
A pilot study to explore and determine feasibility and safety of the administration of surfactant through a new supraglottic device in patients from 500 to 5000 grams with RDS.

DETAILED DESCRIPTION:
Surfactant therapy can be life-saving for newborn infants with respiratory distress due to surfactant insufficiency, also known as respiratory distress syndrome (RDS). All commercially available surfactants for clinical use are approved for administration through an endotracheal tube. Placement of an endotracheal tube, a procedure called intubation, is stressful for the infant and associated with significant adverse effects. The proposed supraglottic instillation device allows infants to benefit from surfactant therapy while avoiding the negative effects of intubation.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at the time of enrollment ≥ 24 0/7 weeks
* Weight at the time of enrollment 500- 5000 grams
* Age ≤ 24 hours old
* Require non-invasive respiratory support (i.e. continuous positive airway pressure, high flow nasal cannula or non-invasive ventilation)
* Require FiO2 ≤ 40%
* Clinical diagnosis of RDS

Exclusion Criteria:

* Prior surfactant administration
* Prior mechanical ventilation
* Major congenital anomaly
* Abnormality of the airway
* Respiratory distress secondary to an etiology other than RDS (suspected pulmonary hypoplasia, pneumothorax, meconium aspiration syndrome, pneumonia, septic or hypovolemia shock, hypoxic ischemic encephalopathy)
* Apgar score < 5 at 5 minutes of age

Min Age: 24 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Estimated)
Dates: Start 2025-02-07 (Estimated); Primary Completion 2025-12-12 (Estimated); Study Completion 2026-03-12 (Estimated)

PRIMARY OUTCOMES:
Instillation failures | First 10 minutes after surfactant instillation.
  Instillation failure is defined as a lack of clinical response
Treatment failure | First 3 days of life
  "Treatment failure" defined as requiring intubation and liquid surfactant instillation with or without mechanical ventilation.

SECONDARY OUTCOMES:
Clinical response | 3 days
  Duration of oxygen therapy
Clinical response | 3 days
  duration of non-invasive respiratory therapy
Clinical response | 3 days
  number of rescue surfactant doses
Clinical response | 3 days
  incidence of pulmonary air leak
Clinical response | 3 days
  pulmonary hemorrhage
Clinical response | defined as need for oxygen at 36 weeks post menstrual age
  chronic lung disease

CONTACTS AND LOCATIONS:
Overall Officials: Kari Roberts, MD, Study Chair — Kari Roberts, MD - University of Minnesota, Minneapolis, MN
Locations (4):
- United States (4):
  - Sharp Mary Birch Hospital for Women & Newborns, San Diego, California
  - Johns Hopkins All Children's Hospital, St. Petersburg, Florida
  - Sisters of Charity Hospital, Buffalo, New York
  - Jackson-Madison County General Hospital, Jackson, Tennessee